CLINICAL TRIAL: NCT07391254
Title: Impact of Omega-3 Supplementation on Omega-3 Status, Vitamin D and Mood in College Students
Brief Title: Omega-3 Supplementation and Mental Health in College Students
Acronym: OMEGA-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Margaret Harris, Associate Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-164
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Mental Health; Vitamin D
Keywords: omega-3; Fish oil; mood; depression; anxiety; mental health; vitamin D; college students; young adults
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The coordinators recruiting and measuring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLacebo (Placebo Comparator): Participants received placebo capsules daily for the duration of the study
  Interventions: Dietary Supplement: Placebo
- Low dose Omega 3 (Experimental): Participants received 700 mg/day of omega 3
  Interventions: Dietary Supplement: Low dose Omega 3
- High dose omega 3 (Experimental): Participants received 2150 mg/day of omega 3 fatty acids
  Interventions: Dietary Supplement: High dose Omega 3

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: PLacebo
Dietary Supplement: Low dose Omega 3 — 700 mg/day omega 3 fatty acids
  Arms: Low dose Omega 3
Dietary Supplement: High dose Omega 3 — 2150 mg/day omega 3 fatty acids
  Arms: High dose omega 3

SUMMARY:
This randomized, placebo-controlled double blinded study examined whether placebo, low- or high dose omega 3 fatty acid supplementation had associations with mental health symptoms and vitamin D status in college students aged 18-27.

DETAILED DESCRIPTION:
A 3-arm randomized design was employed where participants took 2 pills daily for 90 days. The first arm was a placebo, second arm was a low dose omega 3 and third arm was high dose omega 3. Mental health outcomes were measured using the GAD 7 questionnaire that measured anxiety, PHQ-9 which measured depression, and MSQ (Medical Symptoms Questionnaire) that assessed overall bodily symptoms. Vitamin D levels were also assessed as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* age 18-27 years
* if taking antidepressants or enrolled in therapy, needs to be stable with at least 6 months or more of stable medication dose use and regular therapy appointments

Exclusion Criteria:

* age younger than 18 and older than 27
* not willing to take two capsules daily for 90 days
* not willing to get bloodwork
* has a history of fainting during bloodwork
* not willing to have anthropometrics measured
* not willing to have daily text reminders sent to phone
* currently has regularly taken omega 3 daily for at least 6 months
* currently has regularly taken vitamin D supplementation daily for at least 6 months
* allergic or sensitive to fish
* will not like to deal with potential "fish burps"
* utilized mental health services for less than 6 months
* taken an antidepressant for less than 6 months
* currently actively takes benzodiazepines
* currently actively takes sedatives or tranquilizers
* Currently is taking steroid supplements
* currently is taking steroid medications
* had surgery within the last 2 weeks or plans on having surgery within the next 3 months
* currently taking blood thinning medications
* takes NSAIDS regularly
* currently using a weight loss drug

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Anxiety | Baseline to end of intervention (90 days)
  GAD-7
Depression Symptoms | Baseline to end of intervention (90 days)
  PHQ-9

SECONDARY OUTCOMES:
Vitamin D | Baseline to end of intervention (90 days)
  serum 25-hydroxyvitamin D
Medical Symptom Burden | Baseline to end of intervention (90 days)
  Medical Symptoms Questionnaire (MSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Harris, PhD MS HC, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- University of Colorado Colorado Springs, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset, along with the study protocol, statistical analysis plan, informed consent document, and clinical study report, will be made available to qualified researched upon reasonable request. Data will be provided for purposes of research synthesis, including systematic reviews and meta- analyses, following investigator approval and execution of a data use agreement. All shared materials will be de-identified and limited to variables necessary to address the approved research question.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of primary results and within 3 years of that publication.
Access Criteria: Access to de-identified individual participant data will be provided to qualified researchers for the purpose of inclusion in systematic reviews and meta-analyses. Requests must be addressed to the main and backup contacts (Dr Harris and Dr Hutchins) via email (and will be reviewed by the research team). Requests must include a brief research proposal, statistical analysis plan, and evidence of IRB approval or exemption, as applicable. Approved requests will receive the de-identified data and supporting documents via a secure electronic transfer following execution of a data use agreement.